CLINICAL TRIAL: NCT01116531
Title: Efficacy, Safety, Tolerability and Pharmacokinetics of Concomitant Administration of Tramadol With Duloxetine or Pregabalin: a Randomized Controlled Flexible-dose Study in Patients With Neuropathic Pain
Brief Title: Efficacy, Safety, Tolerability and Pharmacokinetics of Concomitant Administration of Tramadol With Duloxetine or Pregabalin
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Helsinki (Other)
Responsible Party: Klaus T Olkkola, MD, Prof, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 60/180/2009
Record Dates: First submitted 2010-04-19; First posted 2010-05-05 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Diabetic Polyneuropathy; Postherpetic Neuralgia
Keywords: Pharmacokinetics; Pharmacodynamics; Interaction; tramadol; duloxetine; pregabalin
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia, Postherpetic | interventions — Tramadol; Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine and tramadol (Active Comparator): To ascertain the double-blinding of subjects and investigators, duloxetine and pregabalin will be administered as 2 similar capsules twice a day. Each of these capsules will contain either 30mg of duloxetine, 75 mg of pregabalin or placebo. Capsules will be prepared at the hospital pharmacy.
  Interventions: Drug: Tramadol; Drug: Duloxetine
- Pregabalin and tramadol (Active Comparator): To ascertain the double-blinding of subjects and investigators, duloxetine and pregabalin will be administered as 2 similar capsules twice a day. Each of these capsules will contain either 30mg of duloxetine, 75 mg of pregabalin or placebo. Capsules will be prepared at the hospital pharmacy.
  Interventions: Drug: Tramadol; Drug: Pregabalin

INTERVENTIONS:
Drug: Tramadol — Initial dose of oral tramadol (depottabl Tramal retard, Orionpharma, Finland) will be 100mg once daily. If the subject is currently on opioid treatment with codeine, tramadol or buprenorphine, the opioid treatment will be stopped, and an equal dose of tramadol will be used as the initial dose. The dose will be titrated on visits V2 and V3 based on the adequacy of pain relief and tolerability. If pain intensity ≥ 4 on a numeric rating scale of 0-10 during V2 and V3 and tramadol is well tolerated, the daily dose will be increased by 100mg. The maximum daily dose of 400 mg tramadol will not be exceeded. If the subject does not tolerate the initial dose of tramadol, he/she will be dropped out of the study and replaced by another patient.
Drug: Duloxetine — The initial dose of duloxetine (Cymbalta, Eli Lilly, USA) will be 30mg once daily. The dose will be titrated on V2 based on the adequacy of pain relief and tolerability. If pain intensity during V2 is < 4 on a scale of 0-10, the dose of duloxetine dose will be 30mg daily throughout the study. If pain intensity is ≥ 4 on a numeric rating scale of 0-10 and duloxetine is well tolerated, the daily dose will be increased to 60mg once daily. If the subject does not tolerate the initial dose of duloxetine, he/she will be dropped out of the study and replaced by another patient.
  Arms: Duloxetine and tramadol
Drug: Pregabalin — The initial dose of pregabalin (Lyrica, Pfizer, USA) will be 75mg twice a day. The dose will be titrated on V2 based on the adequacy of pain relief and tolerability. If pain intensity during V2 is < 4 on a scale of 0-10, the initial dose of pregabalin dose will be continued. If pain intensity is ≥ 4 on a numeric rating scale of 0-10 and pregabalin is well tolerated, the daily dose will be increased to 150mg twice a day. If the subject does not tolerate the initial dose of pregabalin, he/she will be dropped out of the study and replaced by another patient.
  Arms: Pregabalin and tramadol

SUMMARY:
Tramadol is an opioid analgesic, which is widely used in the treatment of acute and neuropathic pain. Treatment of neuropathic pain often requires a combination of pain medications due to the complex nature of neuropathic pain and frequent inadequate response to drug treatment. Common drugs used concomitantly with tramadol are SNRI antidepressant duloxetine and anticonvulsants such as pregabalin. Both tramadol and duloxetine have serotonergic effects and duloxetine has also a potential to inhibit metabolism of tramadol. The objective of the study is to investigate the pharmacokinetics and pharmacodynamic interaction of oral tramadol with duloxetine and pregabalin in patients with chronic neuropathic pain due to postherpetic neuralgia or diabetic polyneuropathy. All subjects will receive tramadol and duloxetine or tramadol and pregabalin in a randomized double-blind order. Primary end point is O-desmethyltramadol concentration.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (≥ 6 months) neuropathic pain due to postherpetic neuralgia or diabetic polyneuropathy
* Pain intensity ≥ 4 on a numerical scale of 0-10
* Informed consent

Exclusion Criteria:

* Clinically significant abnormalities in laboratory screening
* Pregnancy
* Depression
* Use of strong opioids (morphine, oxycodone, fentanyl, hydromorphone, methadone)
* A previous history of intolerance or allergy to the study drugs or to related compounds and additives
* Existing or history of seizures, haematological disorders, clinically significant renal, hepatic, respiratory, cardiac or psychiatric disease, dementia, drug allergy
* Previous or present alcoholism, drug abuse, psychological or other emotional problems or cognitive impairment that are likely to invalidate informed consent or limit the ability of the subject to comply with protocol requirements
* Concomitant drug therapy known to cause significant enzyme induction or inhibition of CYP 1A2, 2D6, 3A4, 2B6, drugs metabolised by CYP2D6 enzyme, antidepressants, MAO-inhibitors, non-steroidal anti-inflammatory analgesics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of O-desmethyltramadol | 3 weeks

SECONDARY OUTCOMES:
Plasma 5-HT concentration | baseline, 1, 2 and 3 weeks
Platelet function | baseline and 3 weeks
Pain intensity | daily for 3 weeks
  Pain intensity will be rated by the subjects on a numerical 11-point rating scale of 0-10 (NRS) with 0 meaning "no pain" and 10 meaning "pain as bad as you can imagine". The subjects will be asked to rate pain intensity on the average over the past 24 hours. Pain intensity will be recorded at each study visit and daily by the subject using a pain diary.
Use of rescue medication | 1,2 and 3 weeks
Behavioral serotonergic effects | 1, 2 and 3 weeks
Concentration of O-desmethyltramadol | baseline, 1 and 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus T Olkkola, MD,PhD,Prof, Principal Investigator — Turku University Hospital and Turku University
Locations (1):
- Department of Anaesthesiology, Intensive Care, Emergency Care and Pain Medicine, Turku University and Turku University Hospital, Turku, Finland